CLINICAL TRIAL: NCT07062796
Title: Access-H20: Sensor-driven Smart Faucet to Enable and Empower Independent Drinking and Grooming for Individuals Impacted by Spinal Cord Injury
Brief Title: Access-H20: Sensor-driven Smart Faucet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Old Dominion University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Anna Jeng, Professor, Old Dominion University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: R44HD108061 (NIH); 2R44HD108061-02 (NIH)
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injury Cervical
Keywords: activities of daily living

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Faucet Water Output Activation (Other): Each SCI subject was instructed to activate the water output modes for drinking and grooming using three different control methods of the faucet: placing their hand near the motion sensor (motion control), using a speech speaker (voice control), and using a remote sensor. For each activity of daily living (drinking and grooming), the physical therapist rated and recorded as "task completed", "partially completed", and "not completed."
  Interventions: Device: Water Faucet

INTERVENTIONS:
Device: Water Faucet — Access H2OTM faucet is a smart, hand free faucet that is designed for ease water access for physical limitations

SUMMARY:
The project's objective was to test the functionality of the upgraded Access H2O faucet prototype designed to support individuals living with spinal cord injury (SCI) for water access for activities of daily living (ADL), including drinking and grooming.

DETAILED DESCRIPTION:
Conventionally, a bathroom faucet includes a hot and cold-water knob used to control flow of water through the faucet, which is utilized for hand washing, face washing, rinsing after brushing, etc. However, existing faucets are inconvenient to use for purposes other than conventional hand washing, unhygienic, and result in wasting large amounts of water. Existing faucets make it difficult for individuals with cervical spinal cord injury (SCI) to carry out basic activities of daily living (ADLs), such as drinking, rinsing their mouths, and washing their faces.

To address these challenges, Nasoni Inc. develop the new faucet, Access H2OTM faucet, to address these challenges. During the Phase I study from 2022-2023, we achieved the following objectives: 1) Successfully designing and producing a prototype of the Access H2O faucet that met input specifications in bench testing, and 2) Developing control algorithms using sensor-based inputs successfully allowed both control and SCI subjects to accurately access desired water. The clinical feasibility study showed that the faucet could improve water access for SCI subjects and improve their ADLs. SCI subjects showed a strong preference for Access-H2O faucets compared to traditional methods.

Before proceeding with commercialization, it is necessary to optimize the operational functions of the prototype. In the Phase II study, the engineering team has planned to enhance the prototype's faucet form factor design and sensors based on the findings from the Phase I study. These enhancements include: 1) optimizing the form factor and nozzle water delivery, 2) refining the sensor & display components, and 3) expanding sensor integration capabilities. Also, the team has improved the water control mechanisms established in Phase I by integrating Access-H2O faucet intelligent algorithms and developing a supporting digital platform with a mobile app & care provider web dashboard to support product efficacy, usability, and field maintenance.

The project's objective was to test the functionality of the upgraded Access H2OTM faucet prototype designed to support individuals living with spinal cord injury (SCI) for water access for activities of daily living (ADL), including drinking and grooming.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with ages 18 to 90 years old are eligible for the study. Individuals should have been screened by a physical or occupational therapist to verify your spinal cord injury (SCI), they are able to follow instructions, they are able to move their eyes and head up, down, and right to activate sensors, and they are able to safely access a bathroom at home.

Exclusion Criteria:

* Individuals have cognitive deficits, mental health, or medical conditions that would keep them from participating in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Water Output Mode Activation | From enrollment to the end of assessment at two days
  Each subject was measured to determine whether she or he can complete the procedures to activate the water output modes (voice, hand motion, and a remote control) of the Access H2O faucet for drinking and grooming. Primary outcomes include "task completed", "task partially completed", and "not completed."

CONTACTS AND LOCATIONS:
Overall Officials: Anna Jeng, ScD, Principal Investigator — Old Dominion University
Locations (1):
- Monarch Physical Therapy Clinic, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
We don't plan to share individual participant raw data; however, aggregated and tabulated data will be published in peer-reviewed articles.